CLINICAL TRIAL: NCT03662828
Title: Epidemiological Description of the Kaposi's Disease in France's Southeast
Acronym: KAPOSI-1
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: KAPOSI-1
Record Dates: First submitted 2018-07-23; First posted 2018-09-10 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-02

CONDITIONS: Kaposi's Disease
Keywords: Kaposi's disease; HHV8; Prevalence
MeSH Terms: conditions — Xeroderma Pigmentosum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the prevalence of the Kaposi's disease in France's southeast on 10 years (from 2007 to 2017)

DETAILED DESCRIPTION:
Kaposi's disease is a multifocal disease with cutaneous expression in more than 95% of cases.

There are 4 forms : Mediterranean, Endemic (Sub-Saharan Africa), iatrogenic and epidemic (HIV) The physiological hypotheses to explain the disease are not clear. A proliferation of immunity cells in blood vessels and also an undetermined role of the human herpes virus 8 (HHV-8) could be involved.

The treatment is complex and not standardized. There are a lot of different treatments.

The purpose of this study is to evaluate the prevalence and described the characteristics and the treatment of the Kaposi's disease in the France's southeast on 10 years, from 2007 to 2017.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed patients with a Kaposi's disease by biopsy from January 2007 to December 2017

Exclusion Criteria:

* Opposition to the use of personal data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed patients with a Kaposi's disease by biopsy from January 2007 to December 2017
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Kaposi's disease | 10 years (2007-2017)
  Diagnosed patients with biopsy, in France's southeast

SECONDARY OUTCOMES:
Descriptive analysis of the different form of the Kaposi's disease in the population | 10 years (2007-2017)
  Mediterranean form, endemic form, iatrogenic form and epidemic form
Descriptive analysis of the population : sociodemographic | 10 years (2007-2017)
  sociodemographic characteristics
Descriptive analysis of the population : paraclinical | 10 years (2007-2017)
  paraclinical characteristics
Descriptive analysis of the population : clinical | 10 years (2007-2017)
  clinical characteristics
Descriptive analysis of the population : therapeutic | 10 years (2007-2017)
  therapeutic care
Survival analysis | 10 years (2007-2017)
  mortality rate

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre Antoine Lacassagne, Nice, Alpes-Maritimes
  - CHU Nice, Nice, Alpes-Maritimes
  - HIA Laveran, Marseille, Bouche Du Rhone
  - CHI de Fréjus, Fréjus, Var
  - Hôpital d'Instruction des Armées Sainte-Anne, Toulon, Var

IPD SHARING:
Plan to Share IPD: No